CLINICAL TRIAL: NCT06345664
Title: Interdisciplinary, E-health Based, Multimodal Follow-up of Somatic, Sleep-related and Psychological Symptoms of Very Immature Preterm Born Babies in Different Age Groups for the Further Development of Previous Care Structures
Brief Title: Interdisciplinary E-health Based Follow-up of Preterm Born Children
Acronym: NeoUp
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, PD Dr. Annette Conzelmann, Principal Investigator, University Hospital Tuebingen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 548/2022BO1
Record Dates: First submitted 2024-02-27; First posted 2024-04-03 (Actual); Last update posted 2025-03-19 (Actual); Status verified 2025-03

CONDITIONS: Preterm Birth
Keywords: preterm born children; ehealth; development; somatic and mental problems; interdisciplinary care
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic assessments and intervention (Other): All families get a diagnostics and intervention recommendations.
  Interventions: Other: Diagnostics and intervention recommendations

INTERVENTIONS:
Other: Diagnostics and intervention recommendations — All families get the same diagnostics and receive individual treatment recommendations.
  Other Names: Differentiated diagnostics and treatment recommendations

SUMMARY:
The aim of the study is to assess mental and somatic symptoms of preterm born children at the ages of 2, 5 and 10 by a multidisciplinary team and to evaluate an app that screens for these symptoms. Furthermore, there will be an evaluation of an intervention by our multidisciplinary team that provides recommendations for further treatment and diagnostic procedures of the children.

DETAILED DESCRIPTION:
* At first, there will be focus groups with experts and affected families to finalize and optimize the study procedure. After that, 90 children will be recruited (ages 2, 5 and 10)
* T0: App-questions for the children at the ages of 5 and 10 and the parents of all children to mental, somatic and sleep problems of the children and well-being of the parents, sleep tracking and recording of a sleep sequence of the children; differentiated examinations and questionnaires to mental and somatic problems of the children by interdisciplinary study team
* Interdisciplinary study team meeting to generate recommendations for the families
* Interdisciplinary study team recommendations for the families
* T1: Comparable to T0 but only measurements that were assessed with questionnaires/at home plus post-experimental questionnaire
* Focus groups with participating families and the study team experts for evaluation of the study procedure and intervention

ELIGIBILITY:
Inclusion Criteria:

* female and male preterm born children (<32 week of pregnancy) that are treated at the clinic in Tübingen and their parents
* Existence of systematical neonatal data and consent of the care person to use this data
* Existence of the data of the 2 year regular follow-up (for the 5 and 10 year olds)

Exclusion Criteria:

* lack of access to a mobile phone/tablet including internet access
* insufficient knowledge of the German language of both parents

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Bayley Scales of Infant and Toddler Development | Baseline
  IQ testing
Wechsler Intelligence Scale for Children (WISC-V) | Baseline
  IQ testing
Children's Sleep Habit Questionnaire (CSHQ-DE 4-10) | Baseline and 36-38 weeks after baseline
  Screening of sleeping behaviour
Sleep Self Report (SSR) | Baseline and 36-38 weeks after baseline
  Screening of sleeping behaviour
Somatics | Baseline and 36-38 weeks after baseline
  Questions to somatic symptoms (diagnoses, inpatient stays, medication, early support) physical therapy, hearing impairment or visual disturbance, pulmonary symptoms, seizure disorders, health related quality of life, body weight, size)
Child Behavior Checklist (CBCL) | Baseline and 36-38 weeks after baseline
  Screening for mental illness
Youth Self Report (YSR) | Baseline and 36-38 weeks after baseline
  Screening for mental illness
Diagnostic-system for mental illness for children and adolescents - III (DISYPS-III SCREEN FBB and SBB) | Baseline and 36-38 weeks after baseline
  Screening for mental illness
KIDSCREEN-27 (The KIDSCREEN) | Baseline and 36-38 weeks after baseline
  Health related quality of life
Parent's Stress Inventory (EBI) | Baseline and 36-38 weeks after baseline
  Load as parents and relationship to the child
App-questions | Baseline and 36-38 weeks after baseline
  Questions reflecting the questionnaires
Postexperimental questionnaire | 36-38 weeks after baseline
  Evaluation of the study

SECONDARY OUTCOMES:
Demographic data | Baseline
  age, gender, ethnicity, perinatal data from previous study participation
Actigraphy measurement | Baseline
  Device that the children are wearing at their wrists
Video of a sleeping sequence | Baseline
  The parents are taking a short video sequence of their sleeping child
Sleep cartoon for children | Baseline and 36-38 weeks after baseline
  Cartoon sleep behavior
Kiddie-Sads-Present and Lifetime Version (K-SADS PL) | Baseline
  Screening mental Illness
Self efficacy dealing with social situations (WIRKSOZ) | Baseline and 36-38 weeks after baseline
  Self-efficacy measurement for social situations in children
Group interviews | Baseline and 36-38 weeks after baseline
  Group interviews with experts and families to get feedback about the study procedure and needs

CONTACTS AND LOCATIONS:
Overall Officials: Annette Conzelmann, Prof. Dr., Principal Investigator — University Hospital Tuebingen; Axel Franz, Prof. Dr., Principal Investigator — University Hospital Tuebingen; Mirja Quante, Dr., Principal Investigator — University Hospital Tuebingen; Ándrea Bevot, Dr., Principal Investigator — University Hospital Tuebingen; Tobias Renner, Prof. Dr., Principal Investigator — University Hospital Tuebingen
Locations (1):
- University Hospital Tuebingen, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: Yes
We share study material and statistical outputs.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Any time before and after completion of the study for 10 years.
Access Criteria: Upon request.